CLINICAL TRIAL: NCT01085643
Title: The Effect of Lubiprostone on Patterns of Contractions in the Small Bowel in Female Patients With Constipation Predominant Irritable Bowel Syndrome (C-IBS)
Brief Title: Effect of Lubiprostone on Small Bowel Contractions in Female Patients With Constipation Irritable Bowel Syndrome (C-IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Edy E Soffer, MD, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 17482
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Results first posted 2011-12-12 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-11

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome
Keywords: IBS; Lubiprostone; Small Bowel; High Resolution Manometry; Delayed Intestinal Transit
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Active Comparator): Same patients are included in both the Lubiprostone arm and the Placebo arm. The reason why the same patients are assigned to two arms is because an effect comparison is done after taking the placebo and later after taking the lubiprostone.
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Same patients are included in both the Lubiprostone arm and the Placebo arm. The reason why the same patients are assigned to two arms is because an effect comparison is done after taking the placebo and later after taking the lubiprostone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 24mcg PO taken once
  Other Names: Amitiza
  Arms: Lubiprostone
Drug: Placebo — 24mcg placebo capsule taken once
  Arms: Placebo

SUMMARY:
Irritable Bowel Syndrome (IBS) is a common disorder, defined by symptom-based diagnostic criteria. The pathogenesis is multifactorial and gut motor dysfunction is considered to be a contributing factor. Changes in motor patterns in the small bowel in IBS patients are quantitative rather than qualitative with no distinct patterns to distinguish patients from healthy individuals. Changes in motor patterns can affect transit of bowel contents. Indeed, variation in intestinal transit was reported in patients with IBS.

Lubiprostone is a novel agent that is Food and Drug Administration (FDA) approved for the treatment of chronic constipation. More recently 2 randomized double-blind, placebo-controlled trials showed the drug to be effective in relieving symptoms in patients with constipation-predominant Irritable Bowel Syndrome (C-IBS), resulting in approval for female patients with C-IBS at a dose of 8 micrograms twice a day.

The investigators hypothesize that lubiprostone works not just as a laxative, but by actually altering motility patterns in the small intestine of female patients with C-IBS. These alterations can be measured through High Resolution Manometry (HRM), a new technique that uses catheters with multiple closely spaced sensors and special software that uses color schemes to portray a pressure gradient. This technique allows a detailed assessment of the direction and spread of contractions. The investigators would like to use HRM to see if lubiprostone affects intestinal contractions by giving blinded participants lubiprostone and placebo while they are undergoing High Resolution Manometry and seeing if any changes in contractions occur. Participants will be recruited from investigator's clinic. If interested, potential subjects will be provided with a copy of the consent form for review. Patients will be informed that after they have had an opportunity to review the consent form, they may contact the study team to further discuss the research and address any questions/concerns they have.

Participants will undergo a screening visit and a manometry visit. During the screening visit investigators will determine eligibility, including application of inclusion/exclusion criteria and administration of a pregnancy test. Then during the manometry visit patients will receive two capsules, lubiprostone and placebo, three hours apart during HRM. Patients will receive each capsule only once and will not know which order they're receiving them in.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a common disorder, defined by symptom-based diagnostic criteria. The pathogenesis is multifactorial, and gut motor dysfunction is considered to be a contributing factor. Dysmotility affects both the small bowel and the colon. Changes in motor patterns in the small bowel in IBS are quantitative rather than qualitative, with no distinct patterns to distinguish patients from healthy individuals. Changes in motor patterns can potentially affect transit of bowel contents and contribute to symptoms. Indeed, variation in intestinal transit was reported in patients with IBS. Small bowel transit studies, using scintigraphy, radio-opaque markers and hydrogen breath test, have shown that transit is delayed in constipation-predominant Irritable Bowel Syndrome (C-IBS) and accelerated in diarrhea-predominant Irritable Bowel Syndrome (D-IBS).

Lubiprostone is a novel agent that has been Food and Drug Administration (FDA) approved for the treatment of adult males and females with chronic constipation. More recently, 2 randomized, double-blind, placebo-controlled trials showed the drug to be effective in relieving symptoms in patients with C-IBS, resulting in approval for female patients with C-IBS, at a dose of 8 micrograms twice a day.

The investigators hypothesize that lubiprostone works not just as a laxative, but by actually altering motility patterns in the small intestine of female C-IBS patients. These alterations could be measured through High Resolution Manometry (HRM), a new technique that uses catheters with multiple, closely spaced sensors, and special software that uses color schemes to portray a pressure gradient. This technique allows a detailed assessment of the direction and spread of individual contractions.

The investigators would like to use HRM to see if lubiprostone affects intestinal contractions. The investigators would like to achieve this by administering blinded participants lubiprostone and placebo while they are undergoing HRM and seeing if any changes in contractions occur. Participants will be recruited both from the investigator's own clinic and by word of mouth. Patients of the investigators will be approached by a member of the research team during a regularly scheduled clinic visit. If interested, potential subjects will be provided with a copy of the consent form for review. Patients will be given ample time to review the consent form with friends, family, and/or other physicians. Patients will be informed that after they have had an opportunity to review the consent form, they may contact the study team to schedule an appointment with one of the co-investigators to further discuss the research and address any questions or concerns the patient may have. Once all the potential subject's issues and concerns have been addressed, and the individual would like to enroll in the study, an investigator or co-investigator will obtain informed consent. Referring physicians will be asked to give their patients the contact information for the study team and the recruitment process will proceed as described above.

Participants will undergo two visits: a screening visit and a manometry visit. During the screening visit we will determine eligibility, including application of inclusion/exclusion criteria and administration of a pregnancy test. Then during the manometry visit, patients will receive the two capsules (lubiprostone and placebo), three hours apart during HRM. Patients will receive each capsule only once, but they will not know which order they're receiving them in.

Patients may receive lubiprostone without participating in the research study. As lubiprostone is FDA approved, the indications would be the same, however, patients receiving the drug under standard of care would not be undergoing the HRM or receiving a placebo capsule. Patients also may not be required to undergo a washout from their standard medication before starting on lubiprostone.

ELIGIBILITY:
Inclusion Criteria:

* Constipation predominant IBS (C-IBS) patients diagnosed on the basis of Rome III criteria
* Females 18 years or older with no operations (except for appendectomy) or medical conditions that can affect small bowel motility
* Ability to comply with the requirements of the entire study
* Patient has given written informed consent to participate and is willing to participate in the entire study
* Patients must not be pregnant or nursing as evidenced by a negative serum pregnancy test taken 7-10 days prior to the manometry. Any female with a positive pregnancy test will be immediately discontinued from the study

Exclusion Criteria:

* Evidence of structural abnormality of the gastrointestinal tract or disease/conditions. These conditions include (but are not limited to): current evidence of history of inflammatory bowel disease (Crohn's disease or ulcerative colitis), active diverticulitis, duodenal ulcer, erosive esophagitis, gastric ulcer, gastroparesis, gastrointestinal malignancy, Barrett's esophagus, gastrointestinal obstruction, carcinoid syndrome, pancreatitis, cholelithiasis, amyloidosis, ileus, progressive systemic sclerosis (scleroderma), anorexia nervosa
* Patients with previous gastrointestinal surgery other than appendectomy or cholecystectomy
* Evidence of cathartic colon or a history of laxative use, that in the investigator's opinion is consistent with severe laxative dependence such that the patient is likely to require or use laxatives during the study
* Patients with clinically diagnosed diarrhea defined as 3 stools/day that are loose or watery in nature
* Psychosis, schizophrenia, mania, severe depression or major psychiatric illness needing pharmacological treatment. Well-compensated depression does not exclude a potential patient. Antidepressant medication is allowed if patient has been on a stable dose for at least the past 3 months
* Any evidence or treatment of malignancy (other than localized basal cell, squamous cell skin cancer or in-situ uterine cervix cancer that has been resected) within the previous five years
* Clinical evidence (including physical examination, laboratory tests and Electrocardiogram) of non-controlled cardiovascular, respiratory, renal, hepatic, hematologic, neurologic, psychiatric diseases or any disease that may interfere with the study
* Existence of surgical or medical conditions that might interfere with the absorption, distribution, metabolism and excretion of the study drug (i.e., gastrectomy, severe renal insufficiency)
* Symptoms of a significant clinical illness in the preceding two weeks prior to the Screening Visit
* Use of any concurrent prohibited medications e.g., drugs that affect Gastrointestinal (GI) motility including lubiprostone, antibiotics (erythromycin), prokinetics, narcotic analgesics, calcium channel blockers, nitroglycerin, and antispasmodics. Patients must not have taken prohibited medications at least 7 days prior to manometry.
* Planned use of drugs or agents 7 days prior to the Screening Visit that affect gastrointestinal motility and/or perceptions including erythromycin
* Use of an investigational drug or participation in an investigational study, within 30 days of the Screening Visit
* Known hypersensitivity to the drug.
* Based on investigator opinion, evidence of alcohol or drug abuse within the past two years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edy E Soffer, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: March 2010 to December 2010 Recruitment place: GI Motility Clinic
Pre-assignment Details: Subjects will have to stop medications affecting small bowel motility 7 days prior to the procedure. Risks expected in this washout period include recurrence of constipation predominant Irritable Bowel Syndrome symptoms- abdominal pain, bloating and constipation. Subjects will be instructed to call the study staff if symptom recurrence occurs.
Groups:
- Placebo Then Lubiprostone: Subjects will receive the two capsules, lubiprostone and placebo, 24 micrograms each, three hours apart during High Resolution Manometry recording. Subjects will receive each capsule only once and will not know which order they're receiving them in, although, placebo capsule has to be given first to avoid a carry over effect of lubiprostone.
Period: Overall Study
Arm/Group | Placebo Then Lubiprostone
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Placebo Then Lubiprostone
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Secondary Outcome: A Change in Length of Spread of Long Distance Propagating Contractions After Placebo.
Description: Pressure waves are considered to represent contractions if the rise in intraluminal pressure is >10mmHg above the baseline. They are considered propagating if they are recorded in more than one channel and occur within a time frame that allowed a minimal velocity of 0.7cm/sec and maximum velocity of 4cm/sec. All contractions, their direction (antegrade, stationary or retrograde) and the length of spread will be determined for each sequence at baseline (after taking Placebo)and within the following 3 hours.
Time Frame: baseline and within the following 3 hours
Population: Considering the fact that this is a pilot study, per protocol a total of 20 subjects should have been recruited; however, due to the limited time and complexity of the study, only 4 subjects completed the study. Due to that fact an analysis of the outcome measures was not submitted, since the results will not provide a meaningful data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo Then Lubiprostone
Number analyzed (Participants) | 0

2. Primary Outcome: A Change in Length of Spread of Antegrade Contractions After Placebo.
Description: as for outcome 1
Time Frame: baseline and within the following 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo Then Lubiprostone
Number analyzed (Participants) | 0

3. Secondary Outcome: A Change in Length of Spread of Retrograde Contractions After Placebo
Description: as for outcome 1
Time Frame: baseline and within the following 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo Then Lubiprostone
Number analyzed (Participants) | 0

4. Primary Outcome: A Change in Length of Spread of Antegrade Contractions After Lubiprostone
Description: as for outcome 1
Time Frame: baseline and within the following 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo Then Lubiprostone
Number analyzed (Participants) | 0

5. Secondary Outcome: A Change in Length of Spread of Long Distance Propagating Contractions After Lubiprostone
Description: Pressure waves are considered to represent contractions if the rise in intraluminal pressure is >10mmHg above the baseline. They are considered propagating if they are recorded in more than one channel and occur within a time frame that allowed a minimal velocity of 0.7cm/sec and maximum velocity of 4cm/sec. All contractions, their direction (antegrade, stationary or retrograde) and the length of spread will be determined for each sequence at baseline (after taking Lubiprostone)and within the following 3 hours.
Time Frame: baseline and within the following 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo Then Lubiprostone
Number analyzed (Participants) | 0

6. Secondary Outcome: A Change in Length of Spread of Retrograde Contractions After Lubiprostone
Description: as for outcome 5
Time Frame: baseline and within the following 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo Then Lubiprostone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Placebo Then Lubiprostone
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Limited time period resulting in recruitment of only 4 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days